CLINICAL TRIAL: NCT02986997
Title: Over 2000 Procedures of Epidural Anesthesia for Percutaneous Nephrolithotomy - a Retrospective Analysis
Brief Title: Over 2000 Epidural Anesthesias for Percutaneous Nephrolithotomy - a Retrospective Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Karolina Dobrońska, MD, Medical University of Warsaw
Other Study IDs: U/1/2016
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Nephrolithiasis; Anesthesia, Local
Keywords: epidural anesthesia; prone position; percutaneous nephrolithotomy
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Percutaneous nephrolithotomy (PNL) is a renal lithiasis treatment. It is usually two staged: it begins in the lithotomy position for ureteral catheter placement and retrograde pyelography and, subsequently, an optimal renal access is obtained in the prone position. In most of the centers, the PNL is done under general anesthesia (GA) that is associated with a risk of complications due to putting an intubated, muscle-relaxed, unconscious patient in a prone position. In our Department the procedure is usually performed under epidural anesthesia. The aim of this study was to evaluate the epidural anesthesia performed for PNL over the last decade in the Medical University of Warsaw Urology Department

DETAILED DESCRIPTION:
Percutaneous nephrolithotomy is a renal lithiasis endoscopic treatment. It is usually two staged: it begins in the lithotomy position for ureteral catheter placement and retrograde pyelography and, subsequently, an optimal renal access is obtained in the prone position. The PNL is usually two staged. It begins in the lithotomy position for cystoscopic placement of ureteral catheter and retrograde pyelography and, subsequently, a patient is placed mainly in the prone position for percutaneous access and stone removal. This position offers more options for puncture.

In most of the centers, the PNL is done under GA, that is associated with a risk of complications due to putting an intubated, muscle-relaxed, unconscious patient in a prone position. Other complications, including blood transfusion, nausea and vomiting or fever, are more often observed after the general then after the regional anesthesia; the cost of general anesthesia is also higher. The regional anesthesia that can be performed independently for the PNL includes spinal, epidural or combined spinal-epidural blocks. A segmental epidural block is better than spinal anesthesia in terms of hemodynamic stability, postoperative analgesia, patient's satisfaction and reduced incidence of postoperative nausea and vomiting. For epidural anesthesia it takes longer to act than for spinal one but it allows avoiding the motor block so the patient can change the position from lithotomy into prone himself with a little assistance. The position of a patient should not be changed rapidly right after the spinal anesthesia has been performed, due to the risk of too high anesthesia level and hemodynamic complications.

The aim of the study was to evaluate the epidural anesthesia performed for PNL over the last decade in the Medical University of Warsaw Urology Department.

ELIGIBILITY:
Inclusion Criteria:

* PNL procedure

Exclusion Criteria:

* no PNL procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have PNL procedure performed in the Urology Department (Medical University of Warsaw) 2005-2015
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
effectiveness of epidural anesthesia for PNL evaluated by a number of participants having this procedure completed | 5 months
  The investigator evaluates whether the procedure could be completely performed under epidural anesthesia

SECONDARY OUTCOMES:
Epidural anesthesia complication rate evaluated by a number of vessel or spinal puncture | 5 months
  The investigator counts all the vessel and spinal punctures done with the Tuohy needle

CONTACTS AND LOCATIONS:
Overall Officials: Karolina Dobronska, MD, Principal Investigator — I Department of Anaesthesiology and Intensive Care
Locations (1):
- Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No